CLINICAL TRIAL: NCT01359553
Title: Comparison Between Intra-articular Ultrasound Imaging, Non-invasive Ultrasound Imaging, Quantitative MRI Imaging, Contrast-enhanced CT Imaging and Arthroscopy for Diagnostics of Knee Osteoarthritis
Brief Title: Clinical Study of Novel Diagnostic Techniques for Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: University of Oulu (Other)
Collaborators: Oulu University Hospital (Other); University of Eastern Finland (Other); Kuopio University Hospital (Other)
Responsible Party: Principal Investigator, Simo Saarakkala, Associate Professor, University of Oulu
Other Study IDs: UltraRusto
Record Dates: First submitted 2011-05-22; First posted 2011-05-24 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Knee Osteoarthritis; Knee Injuries
MeSH Terms: conditions — Osteoarthritis, Knee; Knee Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Knee pain: Group with knee pain problems referred to an arthroscopy.
  Interventions: Other: Intra-articular ultrasound imaging of knee joint during arthroscopy; Other: Non-invasive ultrasound imaging of knee; Other: Quantitative MRI imaging of knee; Other: Contrast-enhanced CT imaging of knee

INTERVENTIONS:
Other: Intra-articular ultrasound imaging of knee joint during arthroscopy
Other: Non-invasive ultrasound imaging of knee
Other: Quantitative MRI imaging of knee
Other: Contrast-enhanced CT imaging of knee

SUMMARY:
The purpose of this study is to clarify the potential of intra-articular ultrasound imaging, non-invasive ultrasound imaging, quantitative MRI imaging, contrast-enhanced CT imaging and arthroscopy for diagnostics of knee osteoarthritis. All methods will be cross-correlated and compared with the arthroscopic findings.

ELIGIBILITY:
Inclusion Criteria:

* Kellgren-Lawrence grade = 1-3 or cartilage defect detected in MRI
* Age >= 20 years

Exclusion Criteria:

* Tumor or inflammation in the knee
* Severe general diseases
* Diabetes

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be selected from those referred to an arthroscopy because of pain symptoms in the knee.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2011-05; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Arthroscopical OA grade | 2014

CONTACTS AND LOCATIONS:
Overall Officials: Simo Saarakkala, Ph.D., Principal Investigator — University of Oulu and Oulu University Hospital; Petri Lehenkari, M.D., Ph.D., Study Director — University of Oulu and Oulu University Hospital; Miika T Nieminen, Ph.D., Study Director — University of Oulu and Oulu University Hospital; Risto Ojala, M.D., Ph.D., Study Director — Oulu University Hospital
Locations (1):
- Oulu University Hospital, Oulu, Finland